CLINICAL TRIAL: NCT01232907
Title: The Effects of L-carnitine on Fatigue in Spinal Cord Injury
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H10-01570
Record Dates: First submitted 2010-10-29; First posted 2010-11-02 (Estimated); Last update posted 2014-10-08 (Estimated); Status verified 2014-10

CONDITIONS: Spinal Cord Injury (SCI)
Keywords: Spinal Cord Injury (SCI)
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Carnitine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- L-Carnitine (Experimental): This study has a single subject design. Each subject acts as its own control. All subjects will go through intervention phase (treatment with L-Carnitine).
  Interventions: Drug: L-Carnitine

INTERVENTIONS:
Drug: L-Carnitine — L-Carnitine, a pharmaceutical product, for the treatment of fatigue in persons with spinal cord injury will be used for this study. L-Carnitine is a nutrient normally obtained in the fat from meat. It promotes fatty acid oxidation of muscle, thereby promoting efficient energy production. Treatment with L-Carnitine has been shown to produce clinically significant improvement in fatigue in persons with multiple sclerosis (MS), cancer, and in aging populations. While the causes of fatigue in persons with SCI may be multifactorial, successful use of L-Carnitine in MS-related fatigue suggests it may have a role in SCI. Standard treatment will entail daily dosages of 1980 milligrams of L-Carnitine (three 330 mg tablets in the morning and three 330 mg tablets in the evening) for 4 weeks.

SUMMARY:
1. Purpose: To explore the use of L-Carnitine, a pharmaceutical product, for the treatment of fatigue in persons with spinal cord injury (SCI).
2. Hypothesis: Similar to previous research in disabled and aging populations, the investigators hypothesize that treatment with L-Carnitine will result in a significant improvement of clinical fatigue in spinal cord injury clients, effecting a decrease on the Fatigue Severity Scale (FSS) of 0.5 points or more. The investigators expect to see an effect after approximately three weeks of treatment.

As secondary outcomes, the investigators expect to see positive changes in the Centre for Epidemiologic Studies Depression Scale (CES-D)and Visual Analogue Fatigue (VAS-F) and Visual Analogue Pain (VAS-P) scores, due to a combination of previously demonstrated effects of L-Carnitine directly on pain and depression, and the effects of the potential decrease in fatigue.

DETAILED DESCRIPTION:
This is a non-concurrent, multiple baseline single subject research design. This pilot study will treat 4 SCI subjects with L-Carnitine, and track the progress of their fatigue prior to, during and following treatment. The target population includes ASIA A, B or C-level SCI subjects at least one year post SCI, with clinically significant fatigue and the ability to provide consent, aged between 19 and 65 years. SCI subjects older than 65 years of age will be excluded due previous research on the effects of L-Carnitine on healthy aging populations. As L-Carnitine has been shown to have positive effects on various effects of aging, these older subjects will be excluded to avoid potentially confounding effects.

Subjects with SCI ASIA A, B or C injuries will be identified from the outpatient list of GF Strong Rehab Centre. Subjects will be initially contacted by letter (letter attached). In addition, recruitment posters will be posted (poster attached). The research coordinator will follow-up by telephone to answer any questions or provide further information about the study, and obtain verbal consent. Given verbal consent, the research coordinator will screen the potential subject for clinically significant fatigue by orally administering the Fatigue Severity Scale. Subjects are required to have an average score of 4 or more on the questions to qualify.

Treatment will consist of the use of 1980 milligrams daily of L-Carnitine over a period of 4 weeks (three 330 mg tablets in the morning and three 330 mg tablets in the evening).

The study is a multiple baseline single subject research design with 4 subjects. Subjects will be randomly assigned to the different baseline lengths.

Subjects will require 4 study visits with interviews. In addition, subjects will be required to complete a daily adverse events log and self-reported bi-weekly outcome measures for the duration of the study. The duration of the study will vary from 10 to 13 weeks.

At least 5 baseline measurements will be taken for each subject prior to the start of treatment with L-Carnitine. Each subsequent subject will have a progressively longer baseline period prior to starting treatment with the final subject having 12 baseline measurements.

The 4 study visits with interview will occur at enrollment (t=0 weeks), at the commencement of L-Carnitine treatment (t=3, 4, 5 or 6 weeks), at the cessation of L-Carnitine treatment (t=7, 8, 9 or 10 weeks), and at the cessation of post-treatment follow-ups (t=10, 11, 12 or 13 weeks).

The interviews will include administration of the Medical Outcomes Study 36-item Short Form (SF-36) and the Brief Pain Inventory (BPI) tools, measurement of weight and Orthostatic Hypotension (OH), and a review of changes in subject's medications and access to medical services prior to starting the study and/or since the last assessment.

The SF-36 and BPI have both been validated in SCI populations. The SF-36 is a widely used measure of health-related quality of life. One of its domains addresses energy & vitality, which would further describe the effects of L-Carnitine on the individual. The BPI measures pain interference, and has been adapted for disabled populations. Its use will further validate the data from the bi-weekly patient self-reports on pain levels, detailed below.

OH is defined as a decrease in systolic blood pressure of 20 mmHg or more, or in diastolic blood pressure of 10 mmHg or more, within 3 minutes of sitting up from a supine position. OH has been shown to be correlated with fatigue. Weight fluctuations may occur due to treatment, as L-Carnitine has been shown to increase muscle mass and muscular energy. If these effects are dramatic in our population, this may be a positive or a negative condition for future treatment of fatigue with L-Carnitine.

During the initial interview only, the following data will also be collected: demographic information (including age, sex, level of education, marital status, vocational status, cause of injury, level of injury, completeness of injury- ASIA impairment classification, and medication list) and the Functional Co-Morbidity Index for Fatigue FCMI-F (including conditions that may contribute to or affect fatigue such as anemia, sleeping disorders, etc) will be recorded. FCMI-F information will be obtained by the PI from chart review, or from the G.F. Strong electronic records, or failing these two, from the subjects' attending physician.

Bi-weekly, subjects will complete the Fatigue Severity Scale (FSS), the Centre for Epidemiologic Studies Depression 10-question Scale (CES-D), the Visual-Analog Scale for Pain (VAS-P), and a patient fatigue self-report scale (Visual-Analog Scale for Fatigue, VAS-F). Measurements will be taken on Mondays and Fridays in the morning. All of these tools have been used by the researchers in previous studies and previously validated in SCI populations. A log documenting adverse effects will be completed daily with treatment. Subjects will be provided with lined paper and an explanatory letter (attached) detailing the requested information for the effects log, which could include provocation, quality, severity, timing and duration of the effect. On days without adverse effects, subjects will log "no adverse effects".

These biweekly evaluations will commence 3, 4, 5 and 6 weeks before L-Carnitine treatment, progress throughout the 4 weeks of treatment, and continue for 3 weeks following cessation of treatment. The research coordinator will contact the subjects by telephone on the established days each week to ensure compliance. All bi-weekly data will be mailed to the research lab at GF Strong within days of completion to remove bias from subsequent data. Subjects will be provided with pre-paid envelopes.

ELIGIBILITY:
Inclusion Criteria:

* Spinal Cord Injury: paraplegia or tetraplegia (ASIA A, B or C)
* More than 1 year since date of injury
* Clinically significant fatigue, determined by a score on the Fatigue Severity Scale greater than or equal to 4
* Between 19 and 65 years of age
* Ability to provide informed consent

Exclusion Criteria:

* Spinal Cord Injury ASIA D, or lack of Spinal Cord Injury
* Acute phase of rehabilitation: less than 1 year since date of injury
* Fatigue Severity Scale score less than 4
* Under 19 years of age or above 65 years of age
* Inability to provide informed consent
* Lack of proficiency in English, specified by an inability to read/understand consent form and complete tools
* Inability to come to GF Strong for 4 separate visits
* On-going treatment with anticoagulants such as warfarin or acenocoumarol
* Pregnancy, lactation or breast feeding
* History of seizures
* Hypothyroidism
* Severe liver or kidney disease
* Other on-going fatigue treatment over the past 6 months
* On-going treatment with L-carnitine
* Lack of stability on pain or depression medication over the past 6 months, determined by history. The subjects will be asked about any changes in pain or depression medications over the past 6 months. If they have had a change in pain or depression medications or started a new pain or depression medication within the past 6 months, they will be excluded from the study. Subjects will be asked about their use of supplements and the indications for the supplements. Again, a change in supplements used for pain or depression in the past 6 months will result in exclusion from the study.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2010-10; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Fatigue Severity Scores (FSS) will be completed by subjects biweekly | starting from 3,4,5, or 6 weeks following initial visit, will continue throughout the 4 weeks of treatment and for 3 weeks following stop of treatment

SECONDARY OUTCOMES:
Fatigue VAS-F will be completed by subjects biweekly | starting from 3,4,5, or 6 weeks following initial visit, will continue throughout the 4 weeks of treatment and for 3 weeks following cessation of treatment
Pain VAS-P will be completed by subjects biweekly | starting from 3,4,5, or 6 weeks following initial visit, will continue throughout the 4 weeks of treatment and for 3 weeks following cessation of treatment
Depression CES-D will be completed by subjects biweekly | starting from 3,4,5, or 6 weeks following initial visit, will continue throughout the 4 weeks of treatment and for 3 weeks following cessation of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Townson, MD, Principal Investigator — University of British Columbia
Locations (1):
- Rehab Research Lab, GF Strong Rehab Centre, 4255 Laurel Street, Vancouver, British Columbia, Canada

REFERENCES:
- See also: Related Info — http://fatiguefunction.icord.org/